CLINICAL TRIAL: NCT00012181
Title: A PHASE I STUDY OF FLAVOPIRIDOL (NSC# 649890; IND# 46211) IN PATIENTS WITH RELAPSED OR REFRACTORY PEDIATRIC SOLID TUMORS OR LYMPHOMAS
Brief Title: Flavopiridol in Treating Children With Relapsed or Refractory Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01854; ADVL0017; CCG-AO972; CDR0000068491; COG-ADVL0017; NCI-A0972; U01CA097452 (NIH)
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Liver Cancer; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Medulloblastoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Recurrent Childhood Visual Pathway Glioma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Recurrent Retinoblastoma; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Recurrent/Refractory Childhood Hodgkin Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Astrocytoma; Familial ependymoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Burkitt Lymphoma; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Neuroblastoma; Osteosarcoma; Retinoblastoma; Wilms Tumor; Recurrence | interventions — alvocidib

ARMS (1):
- Treatment (alvocidib) (Experimental): Patients receive flavopiridol IV over 1 hour on days 1-3. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Other: pharmacological study

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Phase I trial to study the effectiveness of flavopiridol in treating children who have relapsed or refractory solid tumors or lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of flavopiridol in children with relapsed or refractory solid tumors or lymphomas.

II. Determine the toxic effects and pharmacokinetics of this drug in these patients.

III. Determine the antitumor activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive flavopiridol IV over 1 hour on days 1-3. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 to 6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory solid tumor or lymphoma including:

  * Neuroblastoma
  * Osteosarcoma
  * Ewing's sarcoma
  * Rhabdomyosarcoma
  * Wilms tumor
  * CNS tumors
* Histological verification not required for brainstem tumors
* No acute leukemia
* Not eligible for higher priority COG phase I/II study
* Performance status - Karnofsky 50-100% (over age 10)
* Performance status - Lansky 50-100% (age 10 and under)
* At least 2 months
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3 (transfusion independent)
* Hemoglobin at least 8.0 g/dL (transfusion allowed)
* No granulocytopenia, anemia, and/or thrombocytopenia due to bone marrow involvement
* Bilirubin no greater than 1.5 times normal
* SGPT no greater than 5 times normal
* Albumin at least 2 g/dL
* Creatinine no greater than 1.5 times normal
* Creatinine clearance or radioisotope glomerular filtration rate at least lower limit of normal
* Shortening fraction at least 27% by echocardiogram
* Ejection fraction at least 50% by MUGA
* Stable neurologic deficits within the past 2 weeks for patients with CNS tumors
* CNS toxicity less than grade 2
* No active graft-versus-host disease
* No active uncontrolled infection or other serious medical condition
* No uncontrolled diabetes mellitus
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 7 days since prior biologic therapy and recovered
* Prior bone marrow or stem cell transplantation allowed
* At least 6 months since prior allogeneic stem cell transplantation
* At least 1 week since prior growth factors
* No concurrent immunomodulating agents
* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No other concurrent chemotherapy
* Concurrent dexamethasone for CNS tumors allowed if on stable dose for at least 2 weeks prior to study
* Concurrent corticosteroids allowed only for increased intracranial pressure in patients with CNS tumors
* At least 2 weeks since prior local (small port) palliative radiotherapy
* At least 6 months since prior radiotherapy to 50% or more of the pelvis
* At least 6 months since prior craniospinal radiotherapy
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* Recovered from prior radiotherapy
* No concurrent radiotherapy except localized palliative radiotherapy
* No concurrent anticonvulsants

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2001-04; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose at which fewer than one-third of patients experience DLT assessed using Common Toxicity Criteria version 2.0 | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: James Whitlock, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States